CLINICAL TRIAL: NCT06376682
Title: Evaluation of the EPIONE Robotic System for Image-guided Percutaneous Bone Procedures A Prospective Study on Feasibility, Safety and Accuracy
Brief Title: EPIBONE Study: a Prospective Study on Feasibility, Safety and Accuracy
Acronym: EPIBONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Surgical (Industry)
Collaborators: ICUREsearch (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-BO-CIP-0060
Record Dates: First submitted 2024-04-10; First posted 2024-04-19 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Bone Metastases; Fractures, Bone; Bone Tumor
Keywords: Robotic; Robotic guidance; Percutaneous; CT-guided; Bone consolidation; Thermal ablation
MeSH Terms: conditions — Fractures, Bone; Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: The Epione device is an image-guided robotized device that assists the physician during CT-guided procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Patients treated by percutaneous CT-guided procedures in the bone with the EPIONE® device
  Interventions: Procedure: CT-guided bone percutaneous procedure

INTERVENTIONS:
Procedure: CT-guided bone percutaneous procedure — The EPIONE device is a user controlled, stereotactic accessory intended to assist in the planning and manual advancement of one or more instruments, as well as in verification of instrument position during Computed Tomography (CT) guided percutaneous procedures (thermal ablation, bone consolidation, biopsy procedures).

SUMMARY:
Interventional clinical study to obtain performance and safety data of the EPIONE® device when used for bone percutaneous procedures.

DETAILED DESCRIPTION:
The objectives are:

1. To evaluate the feasibility of the Epione robotic assistance for bone percutaneous procedures.
2. To evaluate the safety and the accuracy of the Epione robotic assistance for bone percutaneous procedures.

At least 34 patients (representing at least 67 insertions, as one patient may undergo one or more insertions during the procedure) have been planned for the study. They will be treated by the clinician using the Epione device during a CT-guided percutaneous procedure in musculoskeletal (MSK) structures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years,
2. Patient with indication of CT-guided percutaneous bone procedure under general anaesthesia validated at a multidisciplinary consultation meeting,
3. Patient who has signed an informed consent form,
4. Patient covered by a social security system,

Exclusion Criteria:

1. Patient with contraindication to general anaesthesia,
2. Patient undergoing a procedure without appropriate breathing control,
3. Patient scheduled for CT-guided percutaneous procedures on head and neck, including skull and cervical vertebrae,
4. Patient with medical, psychosocial or emotional conditions unable to fully understand the study protocol, give an uninfluenced informed consent, or meet the study requirements during its whole duration.
5. Pregnant or breast-feeding women,
6. Patient under legal protection (tutorship, guardianship, …),
7. Patient already participating in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste BONNET, Principal Investigator — Gustave Roussy Cancer Institute; Nicolas STACOFFE, Principal Investigator — Hospices Civils de Lyon; Gilles PIANA, Principal Investigator — Paoli-Calmettes Institute
Locations (3):
- France (3):
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred bewteen 16-SEP-2024 and 29-NOV-2024 in the 3 sites. Across the 34 patients included, 90 CT-guided insertions were performed (mean of 2.6 insertions per patient (range: 1-7)).
Units Other Than Participants: Insertion
Period: Overall Study
Arm/Group | Interventional Arm
Started | 34; 90 Insertion
Completed | 32; 84 Insertion
Not Completed | 2; 6 Insertion

BASELINE CHARACTERISTICS:
Units Other Than Participants: Insertion
Groups:
- Interventional Arm: Patients treated by CT-guided percutaneous procedures in the bone with the EPIONE® device
Arm/Group | Interventional Arm
Number analyzed (Participants) | 34
Number analyzed (Insertion) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Patients: Female | 20
  Patients: Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  France | 34
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 24.4 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Successful Introducer Insertion With the EPIONE Device.
Description: To evaluate the feasibility of the EPIONE robotic assistance for bone percutaneous procedures based on a definition of conversion to manual technique
Time Frame: Day of the procedure
Measure: Number; unit: Successful insertion
Units Other Than Participants: Insertions
Arm/Group | Interventional Arm
Number analyzed (Participants) | 34
Number analyzed (Insertions) | 90
Successful insertion | 89

2. Secondary Outcome: Adverse Event(s) (AE)
Description: To evaluate the safety of the EPIONE robotic assistance for bone percutaneous procedures: all AEs (serious and non-serious, related and not-related to the device or the procedure(s))
Time Frame: Up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 34
Participants | 6

3. Secondary Outcome: Lateral Deviation (mm) Accuracy of the EPIONE Robotic Assistance for Bone Percutaneous Procedures
Description: To evaluate the accuracy of the EPIONE robotic assistance for bone percutaneous procedures. Lateral deviation: distance (mm) between the tip of the inserted introducer in its final position and its orthogonal projection on the first planned trajectory
Time Frame: Day of the procedure
Population: Accuracy was measured by insertion. A patient could have multiple introducer insertions during his procedure.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Bone introducer insertions
Arm/Group | Interventional Arm
Number analyzed (Participants) | 34
Number analyzed (Bone introducer insertions) | 90
mm | 2.00 (1.41)

4. Secondary Outcome: Angular Deviation (°)
Description: To evaluate the accuracy of the EPIONE robotic assistance for bone percutaneous procedures. Angular deviation (°): 3D angle between the inserted introducer in its final position and the first planned trajectory.
Time Frame: Day of the procedure
Population: Accuracy was measured by insertion. A patient could have multiple introducer insertions during his procedure.
Measure: Mean (Standard Deviation); unit: °
Units Other Than Participants: Bone introducer insertions
Arm/Group | Interventional Arm
Number analyzed (Participants) | 34
Number analyzed (Bone introducer insertions) | 90
° | 3.06 (2.74)

ADVERSE EVENTS:
Time Frame: Up to 1 month
Description: * AE definitions are based on the ISO 14155:2020
  * AE intensity is based on the standardized Society of Interventional Radiology (SIR) classification.
  * Safety data are reviewed by a Data Safety Monitoring Board (DSMB)
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 2/34
Serious Adverse Events (participants affected / at risk) | 4/34
Other Adverse Events (participants affected / at risk) | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=34)
Clinical deterioration (Musculoskeletal and connective tissue disorders) | 1 (1) — Death at day 9 after the procedure due to cancer progression not related to the procedure, not related to the device.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Life-threatening or disabling event/In-patient or prolonged hospitalization at day 18 after the procedure, not related to the device, not related to the procedure. Recovered event. Resolved at D30
Heart decompensated failure (Cardiac disorders) | 1 (1) — Left-sided heart decompensated failure at day 13 after the procedure, due to probable post chemotherapy systolic dysfunction of the left ventricule. Not related to the procedure, not related to the device. Recovered Event, Resolved at day 17.
Clinical deterioration (Musculoskeletal and connective tissue disorders) | 1 (1) — eterioration in general condition and sudden dyspnea. Patient 's death at day 46 after the procedure due to tumor progression. Not related to the procedure, not related to the device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=34)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Increased right cervical and scapular pain at day 46 after the procedure without deficit in metastatic renal cell carcinoma. Not related to the procedure, not related to the device. Resolved at day 47.
Alteration of general condition, nausea and vomiting (Musculoskeletal and connective tissue disorders) | 1 (1) — The day of the procedure, not related to the procedure, not related to the device. Favorable evolution with symptomatic treatment. Event Resolved at day 4.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute dyspnea at day 30 after the procedure in the context of decompensated heart failure and metastatic breast tumor. Not related to the procedure, not related to the device. Event resolved at the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As mentionned in the protocol: "Prior to submitting the results of this study for publication or presentation, the investigator will have to receive the formal validation by the sponsor on the publication manuscript or presentation. In accordance with generally recognized principles of scientific collaboration, co-authorship with any sponsor personnel will be discussed and mutually agreed upon before submission of a manuscript to a publisher".

DOCUMENTS (2):
  • Study Protocol (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT06376682/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT06376682/SAP_001.pdf